CLINICAL TRIAL: NCT01723267
Title: Automated 3D (SonoAVC) vs 2D Ovarian Follicles Assessment in IVF Cycles: a Randomized Controlled Trial
Brief Title: Automated 3D (SonoAVC) Versus 2D Ovarian Follicles Assessment in IVF Cycles: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, avi ben haroush, Head of Fertility Preservation Service,IVF and Infertility Unit, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: rmcavibh-1
Record Dates: First submitted 2012-07-12; First posted 2012-11-07 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Infertility
Keywords: IVF; 3D ultrasound; SonoAVC; patients in IVF treatment
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3D follicles assessment (Active Comparator): During IVF treatment all ultrasound examinations will use 3D- SonoAVC technology. Timing of hCG injection and oocyte collection will be based on follicle volume and 3D-volume based diameter.
  Interventions: Other: 3D follicles assessment
- 2D follicles assessment (Active Comparator): During IVF treatment all ultrasound examinations will use standard 2D ultrasound. Timing of hCG injection and oocyte collection will be based on follicle diameter.
  Interventions: Other: 2D follicles assessment

INTERVENTIONS:
Other: 3D follicles assessment — 3D ultrasound evaluation in IVF treatment (vs 2D ultrasound)
  Arms: 3D follicles assessment
Other: 2D follicles assessment — 2D ultrasound in IVF treatment (vs 3D ultrasound)
  Arms: 2D follicles assessment

SUMMARY:
Accurate assessment of the size of follicles is important in IVF treatment.Timing of oocyte maturation and subsequent egg collection is largely based on follicle size. An accurate assessment of follicle size and appropriate timing of HCG result in retrieval of more mature oocytes, improved fertilization and higher pregnancy rates. in 3D technology- fter the capturing of a 3D image of an ovary, SonoAVC automatically analyzes the volume dataset, identifies the boundaries of hypoechoic follicles, and provides estimates of their absolute dimensions. These measurements include the largest diameters in three orthogonal planes, the mean follicular diameter (MFD), the volume of the follicle, and the volume-based diameter (d(V)) of the follicle. In the current study the investigators aim to evaluate the use of this automated technique of follicle measurement vs. standard 2D technology on the timing of oocyte maturation and subsequent oocyte retrieval. The investigators speculate that 3D assessment will increase the rate of mature oocyte collection, and eventually will improve other treatment outcomes such as fertilization rate.

DETAILED DESCRIPTION:
Not desired

ELIGIBILITY:
Inclusion Criteria:

* Age:18-39, cycle number 1-4

Exclusion Criteria:

* PCOS
* Endometriosis
* Poor ovarian response
* TESA sperm

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
percentage of matured oocytes | one IVF cycle (within two weeks)

SECONDARY OUTCOMES:
Fertilization rate in ICSI | one IVF cycle/ patient (within two weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Avi Ben-Haroush, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- IVF Unit, Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided